CLINICAL TRIAL: NCT05719181
Title: Effect of Recombinant Human Bone Morphogenetic Protein-2 With an Absorbable Collagen Sponge on Stability of Dental Implant: (Split Mouth Randomized Clinical Trial Study of 6\12\2021 to20\4\2023
Brief Title: Effect of Recombinant Human Bone Morphogenetic Protein-2 With an Absorbable Collagen Sponge on Stability of Dental Implant: (Split Mouth Randomized Clinical Trial Study.
Acronym: rhBMP-2
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Abdullah Ali Abbas, master student, University of Baghdad
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 528622
Record Dates: First submitted 2022-12-07; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Hypertension; Diabetes Mellitus; Blood Disease
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Hematologic Diseases | interventions — Bone Morphogenetic Protein 2

STUDY DESIGN:
Intervention Model Description: two groups; first group with protein , second group without (control)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- control group (Experimental): group consist of 16 patients with no protein application
  Interventions: Biological: rhBMP-2

INTERVENTIONS:
Biological: rhBMP-2 — Recombinant Human Bone Morphogenetic Protein-2 with an Absorbable Collagen Sponge .

SUMMARY:
Effect of Recombinant Human Bone Morphogenetic Protein-2 with an Absorbable Collagen Sponge on Stability of Dental Implant: (Split Mouth Randomized Clinical Trial Study.

DETAILED DESCRIPTION:
The Primary outcome will be measuring the effect of rhBMP- 2/ACS in improving the secondary stability of dental implant by using RFA in comparison to control group.

Secondary outcome association of the effect of other factors (ridge dimension, bone density) on dental implant stability.

ELIGIBILITY:
Inclusion Criteria:

* Patients have good oral hygiene.
* Systemic healthy individuals ,Age more than18 years.
* Healed edentulous area for at least 6 months after tooth extraction (delayed implant protocol).
* Patients have at least two missing teeth in the jaw (canine to 1st molar area) indicated for the dental implant.

Exclusion Criteria:

* Presence of systemic diseases preventing implantation.
* Previous implantation or augmentation of the same region.
* The need for additional bone augmentation procedures (such as maxillary sinus augmentation)
* Partial or total edentulous ridge associated with a severe knife-edge ridge .
* Acute infection or any pathological lesion a the implant site.
* Allergy to one of the materials to be used during operation.
* Pregnancy.
* Radiation therapy, bisphosphonate drugs , Osteoradionecrosis.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-03-18 (Estimated); Study Completion 2023-04-20 (Estimated)

PRIMARY OUTCOMES:
Effect of Recombinant Human Bone Morphogenetic The Primary outcome will be measuring the effect of rhBMP- 2/ACS in improving the secondary stability of dental implant by using RFA in comparison to control group. | At the time of surgery ,all measurment (primary stability) was taken which represented the base line data.
  The topical application of rhBMP-2 in the osteotomy site has an effect through improve secondary stability of the dental implant.

CONTACTS AND LOCATIONS:
Overall Officials: Adbullah Al Abbas, B.D.S, Principal Investigator — University of Baghdad
Locations (1):
- University of Baghdad, Baghdad, Alresafa, Iraq